CLINICAL TRIAL: NCT01929707
Title: A Single-Dose, Dose Escalation, Safety, Tolerability, and Pharmacokinetic Study of LY3050258
Brief Title: A Study of LY3050258 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 14935; I6R-MC-DLAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3050258 (Experimental): Single escalating dose of LY3050258 (2 milligram [mg] up to 200 mg) administered in up to two of two periods.
  Interventions: Drug: LY3050258
- Placebo (Placebo Comparator): Single dose of placebo matching LY3050258 administered in up to one of two periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3050258
  Arms: LY3050258
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and how well the body will handle a single dose of increasing strength of study drug LY3050258. Each participant will receive LY3050258 or placebo once, in each of 2 dosing periods. At least 7 days will pass between doses. This study will last approximately 45 days for each participant. Screening is required within 28 days before the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy postmenopausal females, including Japanese participants
* Have a body mass index (BMI) of 18 to 35 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* An abnormal sitting blood pressure as determined by the investigator
* Any abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, places the participant at an unacceptable risk for study participation
* Current use of statins within the last 3 months prior to dosing
* Current or previous use of anabolic steroids in the preceding 6 months prior to dosing
* Use of dehydroepiandrosterone, other potential over-the-counter (OTC) steroidal supplements, or other nutritional products intended to have weight-reduction and/or performance-enhancing effects within 21 days prior to dosing

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a single-dose, incomplete-crossover, dose-escalation study with minimum 7 days between dosing periods. Each participant received either 2 topical doses of LY3050258 or 1 topical dose each of LY3050258 and placebo. Two discontinued participants completing Period 1 were replaced in Period 2.
Groups:
- 2 mg LY3050258 (Trunk): Period 1: Healthy participants received a topical application of 2 milligrams (mg) LY3050258.
- 6 mg LY3050258 (Trunk): Period 1: Healthy participants received a topical application of 6 mg LY3050258.
- 20 mg LY3050258 (Trunk): Period 1: Healthy participants received a topical application of 20 mg LY3050258
- Placebo (Trunk): Period 1 or 2: Healthy participants received a topical application of placebo.
- 60 mg LY3050258 (Trunk): Period 2: Healthy participants received a topical application of 60 mg LY3050258.
- 200 mg LY3050258 (Trunk): Period 2: Healthy participants received a topical application of 200 mg LY3050258.
- 20 mg LY3050258 (Axilla): Period 2: Healthy participants received a topical application of 20 mg LY3050258.
- Placebo (Axilla): Period 2: Healthy participants received a topical application of placebo.
Period: Intervention Period 1
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | Placebo (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla) | Placebo (Axilla)
Started | 6 | 8 | 12 | 10 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 6 | 8 | 12 | 10 | 0 | 0 | 0 | 0
Completed | 6 | 8 | 12 | 7 (Two discontinued participants were replaced in Period 2) | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Washout Period ≥7 Days
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | Placebo (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla) | Placebo (Axilla)
Started | 6 | 8 | 12 | 7 | 0 | 0 | 0 | 0
Completed | 6 | 8 | 12 | 7 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | Placebo (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla) | Placebo (Axilla)
Started | 0 (Incomplete-crossover design) | 0 (Incomplete-crossover design) | 0 (Incomplete-crossover design) | 5 (Incomplete-crossover design) | 6 (Incomplete-crossover design) | 8 (Incomplete-crossover design) | 12 (Incomplete-crossover design) | 4 (Incomplete-crossover design)
Completed | 0 | 0 | 0 | 5 | 6 | 6 | 12 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug
Groups:
- LY3050258 or Placebo: Participants received doses of 2, 6, or 20 mg LY3050258 or placebo during Period 1 by topical administration on the trunk. Participants received 60, 200 mg LY3050258 or placebo on the trunk or 20 mg LY3050258 or placebo by topical administration on the axilla during Period 2. There were at least 7 days between treatments.
Arm/Group | LY3050258 or Placebo
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs which were considered to be related to study treatment by the investigator while on treatment and during the follow-up. Summaries of SAEs and other non-serious adverse events (AEs), regardless of causality, are located in the Reported Adverse Events module.
Time Frame: Baseline up to 21 days postdose
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 2 mg LY3050258 (Trunk): Period 1: Healthy participants received a topical application of 2 mg LY3050258.
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | Placebo (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla) | Placebo (Axilla)
Number analyzed (Participants) | 6 | 8 | 12 | 15 | 6 | 8 | 12 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3050258
Time Frame: Period 1: Predose, 2, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours (h) postdose and Day 7 postdose; Period 2: Predose, 2, 4, 6, 8, 10, 12, 18, 24, 36 and 48 h postdose and Days 7, 14, and 21 postdose.
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data to calculate Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla)
Number analyzed (Participants) | 3 | 8 | 12 | 6 | 8 | 12
nanograms/milliliter (ng/mL) | 0.0397 (81) | 0.0626 (47) | 0.968 (746) | 0.681 (75) | 1.77 (26) | 0.630 (52)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY3050258
Time Frame: Period 1: Predose, 2, 4, 6, 8, 10, 12, 18, 24, 36 and 48 h postdose and Day 7 postdose; Period 2: predose, 2, 4, 6, 8, 10, 12, 18, 24, 36 and 48 h postdose and Days 7, 14, and 21 postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data to calculate AUC(0-∞). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla)
Number analyzed (Participants) | 3 | 6 | 12 | 6 | 8 | 12
nanograms*hour per milliliter (ng*hr/mL) | 1.60 (95) | 7.02 (161) | 17.5 (198) | 41.6 (81) | 88.5 (35) | 23.0 (37)

ADVERSE EVENTS:
Arm/Group | 2 mg LY3050258 (Trunk) | 6 mg LY3050258 (Trunk) | 20 mg LY3050258 (Trunk) | 20 mg LY3050258 (Axilla) | 60 mg LY3050258 (Trunk) | 200 mg LY3050258 (Trunk) | Placebo (Trunk) | Placebo (Axilla)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/12 | 0/12 | 0/6 | 0/8 | 0/15 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 1/12 | 1/12 | 0/6 | 1/8 | 1/15 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY3050258 (Trunk) (N=6) | 6 mg LY3050258 (Trunk) (N=8) | 20 mg LY3050258 (Trunk) (N=12) | 20 mg LY3050258 (Axilla) (N=12) | 60 mg LY3050258 (Trunk) (N=6) | 200 mg LY3050258 (Trunk) (N=8) | Placebo (Trunk) (N=15) | Placebo (Axilla) (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days